CLINICAL TRIAL: NCT01011725
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Efficacy of MK0773 in Healthy Postmenopausal Women
Brief Title: Safety, Tolerability and Efficacy of MK0773 in Healthy Postmenopausal Women (0773-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0773-003; MK0773-003
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — 3-fluoro-N-(3H-imidazo(4,5-b)pyridin-2-ylmethyl)-1,4a,6a-trimethyl-2-oxo-2,4a,4b,5,6,6a,7,8,9,9a,9b,10,11,11a-tetradecahydro-1H-indeno(5,4-f)quinoline-7-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postmenopausal Women- Active Agent Group (Experimental)
  Interventions: Drug: MK 0773
- Postmenopausal Women- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK 0773 — 25 mg oral tablet b.i.d. MK 0773 or 100 mg oral tablet b.i.d. MK 0773, for 12 weeks
  Arms: Postmenopausal Women- Active Agent Group
Drug: Placebo — Placebo oral tablet b.i.d for 12 weeks
  Arms: Postmenopausal Women- Placebo

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, and pharmacodynamic efficacy of MK0773 in healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a nonsurgical postmenopausal female
* Subject is neither grossly overweight nor underweight for her height
* Subject is in good health
* Subject is willing to avoid excess alcohol and strenuous physical activity during the study
* Subject agrees to refrain from consuming St. John's Wort, grapefruit or grapefruit juice during the study

Exclusion Criteria:

* Subject has significant drug allergies
* Subject has donated blood or taken an investigational drug in another clinical trial within the last 4 weeks
* Subject is a regular user or past abuser of any illicit drug (including alcohol)
* Subject drinks excessive amounts of caffeinated beverages
* Subject has a history of cancer

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-11; Primary Completion 2006-04 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious Clinical Adverse Events | From date of enrollment through 12 weeks of study
Number of Participants with Nonerserious Clinical Adverse Events | From date of enrollment through 12 weeks of study
Number of Participants with Serious Laboratory Adverse Events | From date of enrollment through 12 weeks of study
Number of Participants with Nonserious Laboratory Adverse Events | From date of enrollment through 12 weeks of study
Number of Participants Who Discontinued Due to Any Adverse Event | From date of enrollment through 12 weeks of study
Number of Participants Who Withdrew Consent and Discontinued the Study | From date of enrollment through 12 weeks of study
Least Squares Mean Change in Lean Body Mass | From baseline, at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC